CLINICAL TRIAL: NCT05178199
Title: The Effectiveness of "Remote Psychological Support Group" Intervention for Nurses During the COVID-19 Outbreak
Brief Title: The Effectiveness of RPSG Intervention for Nurses During the COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202107077RINC
Record Dates: First submitted 2021-11-15; First posted 2022-01-05 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: psychological support group; nurse; COVID-19; quality of life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Psychological Support Group (Experimental): The study will invite nurses through QR code on line, and assess their background, self-efficacy, fear of COVID-19, psychological distress, and quality of life by questionnaires first. Then four evacuation acute wards (A, B, C, and D) will be randomly allocated, and the two wards will be drawn out as experimental group ward. Each group will be followed for 2 months and their outcomes will be assessed at 3 time points: baseline (pre-RPSG) (T0), and 4 (T1), 8 (T2) weeks after-RPSG, T0-T2, respectively.
  Interventions: Behavioral: RPSG; Behavioral: AVMBM
- Mindfulness through audio and video (Active Comparator): The study will invite nurses through QR code on line, and assess their background, self-efficacy, fear of COVID-19, psychological distress, and quality of life by questionnaires first. Then four evacuation acute wards (A, B, C, and D) will be randomly allocated, and the two wards will be drawn out as experimental group ward. Each group will be followed for 2 months and their outcomes will be assessed at 3 time points: baseline (pre-RPSG) (T0), and 4 (T1), 8 (T2) weeks after-RPSG, T0-T2, respectively.
  Interventions: Behavioral: RPSG; Behavioral: AVMBM

INTERVENTIONS:
Behavioral: RPSG — The RPSG program include sharing successful experience, progressive muscle relaxation (PMR), and mindfulness-based stress reduction (MBSR). The duration is at last 8 weeks and includes 1 hour per week of RPSG activities.
Behavioral: AVMBM — The duration is also at last 8 weeks and includes encouraging to use "5 minutes Audio and Video Mindfulness of Breathing Meditation (AVMBM)" per week.

SUMMARY:
The cases of COVID-19 are continuing to be confirmed around the world. In the clinical settings, the nurses in evacuation acute wards are main responsibility to undertake the care of emergency patient follow-up and suspected or confirmed COVID-19 cases. Those nurses have to face the high psychological pressure, unknown panic, fear and so on. Thus, the study plans to invite nurses who are working in evacuation acute wards to participate the project called "Remote Psychological Support Group (RPSG)". The study supposes "RPSG" could improve nurses' self-efficacy, fear of COVID-19, psychological distress, and quality of life.

DETAILED DESCRIPTION:
The cases of COVID-19 are continuing to be confirmed around the world. In the clinical settings, the nurses in evacuation acute wards are main responsibility to undertake the care of emergency patient follow-up and suspected or confirmed COVID-19 cases. Those nurses have to face the high psychological pressure, unknown panic, fear and so on. Thus, the study plans to invite nurses who are working in evacuation acute wards to participate the project called "Remote Psychological Support Group (RPSG)". The results of this study will establish the effectiveness of RPSG intervention for nurses on self-efficacy, fear of COVID-19, psychological distress, and quality of life and identify the feasibility of the RPSG. The results are also critical to improving the quality of care for nurses during the COVID-19 outbreak and the RPSG model will establish an important basis for support group in the event of other Severe Pneumonia with Novel Pathogens in the future.

ELIGIBILITY:
Inclusion Criteria:

* The nurses have to above 20 years old.
* The nurses who work in evacuation acute wards.

Exclusion Criteria:

* The nurses who have any mental illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
compare self-efficacy of nurses before and after RPSG | 8 weeks
  The study uses structured questionnaires "General Self-Efficacy Scale (GSES)" to evaluate the effectiveness of RPSG. This scale is a self-report measure of self-efficacy, and it includes ten questions, each question score from 1 to 4. The total score is calculated by finding the sum of the all items, and ranges between 10 and 40, with a higher score indicating more self-efficacy.
compare fear of COVID-19 for nurses before and after RPSG | 8 weeks
  The study uses structured questionnaires "the Fear of COVID-19 Scale" to evaluate the effectiveness of RPSG. The Fear of COVID-19 Scale is a seven-item scale with using a five-item Likert-type scale. A total score is calculated by adding up each item score (ranging from 7 to 35). The higher the score, the greater the fear of cororonavirus-19.
compare psychological distress for nurses before and after RPSG | 8 weeks
  The study uses structured questionnaires "distress thermometer (DT) " to evaluate the effectiveness of RPSG. The distress thermometer (DT) is a rating scale used to measure distress: 0 (no distress) to 10 (extreme distress).
compare quality of life for nurses before and after RPSG | 8 weeks
  The study uses structured questionnaires "WHOQOL-BREF Taiwan version" to evaluate the effectiveness of RPSG. The WHOQOL-BREF Taiwan version contains 28 items classified into the same four domains as the standard WHOQOL-BREF, and using a five-item Likert-type scale. A total score of each domain ranging from 4 to 20, with a higher score indicating better quality of life.

SECONDARY OUTCOMES:
satisfaction for RPSG | 8 weeks
  Finally, the study uses Numerical Rating Scale (VRS) to evaluate satisfaction about RPSG for nurses. The scores from zero to ten, the higher scores represent more satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Hsuan Wen, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan